CLINICAL TRIAL: NCT05659602
Title: A Clinical Study to Assess Preliminary Efficacy, Safety and Tolerability of HH-120 Nasal Spray in Participants Diagnosed With Asymptomatic or Mild COVID-19
Brief Title: A Clinical Study to Assess Preliminary Efficacy, Safety and Tolerability of HH-120 Nasal Spray in COVID-19 Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Ditan Hospital (Other)
Responsible Party: Principal Investigator, Ronghua Jin, Chief Physician, Beijing Ditan Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HH120-IIT-NS05
Record Dates: First submitted 2022-12-20; First posted 2022-12-21 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Coronavirus Disease 2019(COVID-19)
Keywords: COVID-19; Treatment
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HH-120 group (Experimental): HH-120 Nasal Spray
  Interventions: Biological: HH-120 Nasal Spray

INTERVENTIONS:
Biological: HH-120 Nasal Spray — HH-120 Nasal Spray 8-10 times per day for 6 consecutive days

SUMMARY:
To evaluate the preliminary efficacy and safety of HH-120 nasal spray in the treatment of asymptomatic or mild COVID-19.

DETAILED DESCRIPTION:
During this study, participants will receive HH-120 nasal spray treatment for 6 consecutive days, the efficacy and safety of HH-120 will be assessed throughout the study period based on viral clearance, clinical recovery, illness severity and adverse events.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 65 years old.
* Participants with mild COVID-19 with symptom onset≤5 days or asymptomatic COVID-19.
* Participants being able and willing to provide informed consent prior to any study-specific procedure.

Exclusion Criteria:

* Participants with moderate or severe COVID-19.
* Participants within the pregnancy or breastfeeding period or plan to be pregnant during the study period.
* Participants requiring oxygen treatment (such as non-invasive ventilation, invasive mechanical ventilation, ECMO, etc.).
* Participants with nasal disease that is inconvenient or intolerant of nasal spray administration, or cannot use the nasal spray treatment.
* Participants with comorbid Malignancy or with a history of malignancy.
* Participants with active or uncontrolled systemic autoimmune disease.
* Insufficient function of key organs.
* Other reasons considered by the investigator to be unsuitable for the trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2022-07-09 (Actual); Primary Completion 2023-01-03 (Actual); Study Completion 2023-01-03 (Actual)

PRIMARY OUTCOMES:
Time to achieving SARS-CoV-2 clearance (defined as negative quantitative Real-Time polymerase chain reaction [qRT-PCR] tests taken on two consecutive days). | Up to 12 days
  Median time from first dose to achieving SARS-COV-2 clearance.
Proportion of participants with SARS-CoV-2 clearance. | Up to 12 days
  Proportion of participants achieving SARS-CoV-2 clearance from the first dose until Day 12.

SECONDARY OUTCOMES:
Clinical recovery of COVID-19. | Up to 12 days
  Time to sustained COVID-19 symptoms recovery; Time to COVID-19 symptoms improvement; Proportion of participants with sustained COVID-19 symptoms recovery; Proportion of participants with COVID-19 symptoms improvement.
Viral load. | Up to 12 days
  Change of CT values of N gene and ORF1 gene (qRT-PCR) from baseline.
Adverse event. | Up to 12 days
  Incidence and severity of adverse events.

OTHER OUTCOMES:
Proportion of the participants who have progression of COVID-19. | Up to 12 days
  Proportion of participants who progress to moderate/severe/critical type of COVID-19 illness.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Ditan Hospital, Capital Medical University, Beijing, Beijing Municipality, China